CLINICAL TRIAL: NCT03889652
Title: Comparison Between OCT Nerve Fiber Layer and Ganglion Cell Complex Parameters Following Cataract Extraction in Patients With or Without Primary Open Angle Glaucoma
Brief Title: Optical Coherence Tomography of Nerve Fiber Layer and Ganglion Cell Complex After Cataract Extraction
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hebatalla Makled, Ophthalmology lecturer, Kasr El Aini Hospital
Other Study IDs: N-68-2018
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cataract; Primary Open-angle Glaucoma
Keywords: Retinal nerve fiber layer (RNFL); Ganglion cell complex (GCC); Optical coherence tomography (OCT); Primary open angle glaucoma (POAG); Cataract
MeSH Terms: conditions — Cataract; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cataract group: Group 1 includes patients who are planned for cataract extraction without any other preexisting retinal or optic nerve pathology that may affect the RNFL thickness.
  OCT (investigation) before and after cataract extraction
  Interventions: Diagnostic Test: Oct scans
- Combined cataract and glaucoma group: Group 2 includes patients who are diagnosed with POAG controlled on medical treatment and have cataract and planned for cataract extraction only OCT is done before and after cataract extraction
  Interventions: Diagnostic Test: Oct scans

INTERVENTIONS:
Diagnostic Test: Oct scans — Oct scans to assess thickness of RNFL and GCC before and after cataract extraction surgery in both groups

SUMMARY:
Optical coherence tomography (OCT) for retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) is done before and after cataract extraction in patients with or without primary open angle glaucoma (POAG)

DETAILED DESCRIPTION:
The investigator's study includes two groups of patients, each consists of 25 eyes, group 1 (cataract group)includes patients who are planned for cataract extraction without any other preexisting retinal or optic nerve pathology that may affect the RNFL thickness, while group 2 (combined cataract and glaucoma group) includes patients who are diagnosed with POAG controlled on medical treatment with cataract and planned for cataract extraction only.

The OCT scans with complete ophthalmological examination are done before surgery and 6 weeks after uneventful cataract extraction (phacoemulsification with intraocular lens implantation)

ELIGIBILITY:
Inclusion Criteria:

• patients with cataract without any other concomitant retinal, optic nerve head pathology other than POAG are included in the study and divided onto two groups

Exclusion Criteria:

* Patients having any retinal or optic nerve pathology that might have affected nerve fiber layer thickness other than POAG eg: high myopia
* POAG patients who are planned for combined surgery
* Refractive errors greater than spherical equivalent of 6 diopters (myopia or hypermetropia)
* Dense cataract hindering OCT imaging
* History of previous ocular surgery or trauma

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cataract without any other concomitant retinal, optic nerve head pathology other than POAG are included in the study and divided into two groups Group 1 patients with cataract only Group 2 patients with cataract and POAG who are planned for cataract surgery only and controlled on medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
RNFL and GCC thickness | Oct scans before and 6 weeks after surgery
  Assessment of RNFL and GCC thickness change after cataract extraction

SECONDARY OUTCOMES:
Final best corrected visual acuity (BCVA) | Six weeks after cataract surgery
  Assessment of the final BCVA recorded according to the Snellen chart and converted to logMAR for statistical analysis

OTHER OUTCOMES:
Intraocular pressure (IOP) change and central foveal thickness (CFT) change | Six weeks after cataract surgery
  Assessment of the IOP and CFT change after cataract extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al-Ainy teaching hospital, Cairo, Egypt